CLINICAL TRIAL: NCT06729697
Title: Pharmaceutical Literacy in Spanish Population and Association With Health-Related Quality of Life
Brief Title: Pharmaceutical Literacy and Quality of Life in Spanish Population.
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Barcelona (Other)
Collaborators: Sociedad Espanola de Farmacia Clinica, Familiar y Comunitaria (Other)
Responsible Party: Principal Investigator, Pilar Modamio, Full Professor, University of Barcelona
Other Study IDs: CER052416
Record Dates: First submitted 2024-11-21; First posted 2024-12-11 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Health Related Quality of Life; Literacy
Keywords: Pharmaceutical literacy; Health related quality of life; Spain; Community pharmacist
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this study is to learn about the knowledge and abilities that patients have regarding their own medication and to see if that's related to their quality of life.

The main questions it aims to answer are:

* Are patients abilities and knowledge about their medications sufficient to ensure a safe and efective use?
* Are those knowledge and abilities related to the patient's quality of life? How?

Patients already taking at least one medication will answer questions about their abilities and knowledge towards medication and their quality of life related to their health state.

DETAILED DESCRIPTION:
A cross-sectional study is carried out, consisting of an interview between the patients and community pharmacists included in the study.

The participants selected are adults usually taking medication that answer questions related to their pharmaceutical literacy (RALPH interview). This type of literacy refers to three domains regarding functional, comunicative and critical abilities about their own medication.

After that, every participant answers a simple survey regarding their health-related quality of life including topics such as mobility, self-care, everyday activities, pain and mental health (EQ-5D-5L survey).

The recruitment and interviewing take place at the same time, and it requires less than 30 minutes per patient. No follow-up is needed afterward.

There are no risks associated with this procedure, and the participation of the patients will always be voluntary and anonymous.

Previously to the patients' enrollment in the study, proper information will be given to the potential participants and an informed consent will be signed.

ELIGIBILITY:
Inclusion Criteria:

* Adults currently taking at least one medication prescribed by a physician and living in Spain.

Exclusion Criteria:

* Having physical or cognitive limitations that make it impossible to answer the study questions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults taking at least one medication in Spain at the moment of the study.
Sampling Method: Non-Probability Sample
Enrollment: 1246 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Recognising and Addressing Limited Pharmaceutical Literacy (RALPH) interview guide score | Through study completion, an average of 1 year.
  A quantitative score will be obtained after an interview using the RALPH guide for community pharmacy. Only correct answered questions will add a point to the score. The values obtained stand between 0 and 10, and a higher score means a better outcome.
EQ-5D-5L index score | Through study completion, an average of 1 year.
  A health state index score will be calculated from individual health profiles using the Spanish value set (Roudijk B, Ludwig K, Devlin N, Roudijk B, Ludwig K, Devlin N. EQ-5D-5L Value Set Summaries. Value Sets for EQ-5D-5L. 2022;55-212.) where the values stand between -0.166 and 1, and a higher score means a better outcome.

SECONDARY OUTCOMES:
Sex | Through study completion, an average of 1 year.
  Sex according to the categories: male or female.
Age | Through study completion, an average of 1 year.
  Age in years.
Country of birth | Through study completion, an average of 1 year.
  Name of the country of birth.
Level of education | Through study completion, an average of 1 year.
  Education level according to the 4 categories: uneducated, primary education, secondary education and higher education.
Situation related to economic activity | Through study completion, an average of 1 year.
  Economic activity according to the 7 categories: working, unemployed, retired, studying, unable to work, mainly engaged in housework and other situations.
Working time | Through study completion, an average of 1 year.
  If working, type of working time according to the categories: full time and part time.
Time since the prescription of the medicine | Through study completion, an average of 1 year.
  Time in months.
Total number of medicines prescribed per day | Through study completion, an average of 1 year.
  Number of medicines prescribed per day according to the categories: less than 5 medicines and more than 5.

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Modamio Charles, PhD, Study Director — University of Barcelona
Locations (1):
- Clinical Pharmacy and Pharmaceutical Care Unit., Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Acording to the protocol aproved by the Bioethics Commission of the University of Barcelona, the IPD will not be shared with other researchers since it is not an interventional study.

REFERENCES:
- [Background] Roudijk B, Ludwig K, Devlin N. EQ-5D-5L Value Set Summaries. 2022 Mar 24. In: Devlin N, Roudijk B, Ludwig K, editors. Value Sets for EQ-5D-5L: A Compendium, Comparative Review & User Guide [Internet]. Cham (CH): Springer; 2022. Chapter 4. Available from http://www.ncbi.nlm.nih.gov/books/NBK589305/ PMID 36810042
- [Background] Andreu-March M, Aguas Compaired M, Marino EL, Modamio P. Cross-cultural adaptation and validation of the Recognizing And Addressing Limited Pharmaceutical Literacy (RALPH) interview guide in community pharmacies. Res Social Adm Pharm. 2023 Jun;19(6):882-888. doi: 10.1016/j.sapharm.2023.02.004. Epub 2023 Feb 16. PMID 36868912